CLINICAL TRIAL: NCT06866548
Title: Safety and Efficacy Evaluation of Anti IGF-1R Monoclonal Antibody Combined With Anti-PD-1 Monoclonal Antibody in Treatment in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Ren Shancheng, Professor, Chief of Urology, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELIX-25
Record Dates: First submitted 2025-03-03; First posted 2025-03-10 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: mCRPC
Keywords: Prostate Cancer; Metastasis; PD-1; IGF-1R
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Insulin-Like Growth Factor I, Resistance To | interventions — teprotumumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with anti-IGF-1R mAb(Teprotumumab/IBI311) + anti-PD-1 mAb (Tislelizumab) (Experimental)
  Interventions: Drug: anti-IGF-1R mAb (Teprotumumab/IBI311) + anti-PD-1 mAb (Tislelizumab)

INTERVENTIONS:
Drug: anti-IGF-1R mAb (Teprotumumab/IBI311) + anti-PD-1 mAb (Tislelizumab) — Drug: Teprotumumab/IBI311 Given by IV infusion Initiate dosing with 10 mg/kg for first infusion, followed by 20 mg/kg every 3 weeks.
  Drug: Tislelizumab Given by IV infusion 200 mg every 3 weeks

SUMMARY:
This trial is designed to evaluate the safety and efficacy of anti-IGF-1R mAb in combination with anti-PD-1 mAb in patients with mCRPC.

DETAILED DESCRIPTION:
This trial is designed to primarily confirm the safety and tolerability of anti-IGF-1R mAb (Teprotumumab/IBI311) in combination with anti-PD-1 mAb (Tislelizumab) using the recommended dose level for patients with mCRPC patients. Additionally，this trial is aimed to evaluate the clinical efficacy of anti-IGF-1R mAb combined with anti-PD-1 mAb in the treatment of mCRPC patients and to investigate whether the combined treatment can enhance endocrine therapy sensitivity in mCRPC patients. As for exploratory objectives，the trial is designed to identify and validate predictive biomarkers associated with therapeutic efficacy and safety profiles of the combination regimen in mCRPC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men over 18 years old and under 85 years old;
2. Diagnosed with prostate adenocarcinoma by prostate biopsy pathology report;
3. Patients with metastatic castration-resistant prostate adenocarcinoma (mCRPC);
4. evidence of metastatic bone lesions on imaging such as PSMA-PET-CT or bone metastasis imaging ECT;
5. Serum testosterone in the depot range (< 50 ng/dL or 1.75 nmol/L);
6. Patients need to be willing to undergo pre- and on-treatment biopsy;
7. ECOG score ≤ 2;
8. Expected survival time of 6 months or more;
9. Substantially normal bone marrow, liver and kidney function:

   1. white blood cell (WBC) > 3 x 10^9 cells/L
   2. Absolute neutrophil count (ANC) > 1×10^9 cells/L
   3. Hemoglobin >9.0 g/dL
   4. Platelet count >100×10^9/L
   5. Serum creatinine <1.5 × upper limit of normal (ULN)
   6. Serum total bilirubin <1.5 × ULN
   7. Serum glutamine aminotransferase <3 × ULN
   8. Aspartate aminotransferase <3 × ULN
10. willingness to cooperate and complete study follow-up and related tests.
11. The subject or his/her representative voluntarily participates in the study and signs a written informed consent; and
12. The questionnaire can be completed in Chinese.
13. The patient has been informed of the trial;

Exclusion Criteria:

1. Histologically predominantly other types of prostate cancer, such as sarcomas, lymphomas, small cell tumors, and neuroendocrine tumors;
2. Active infection requiring parenteral antibiotic therapy or causing fever (temperature > 100.5 o F or 38.1 o C) within 1 week prior to enrollment;
3. have received systemic, ongoing immunosuppressive therapy within 14 days prior to receiving study treatment (except for adrenal replacement steroid doses not exceeding 10 mg prednisone equivalent per day in the absence of active autoimmune disease or short-term steroid therapy (<5 days) within 7 days prior to initiation of study treatment);
4. Subjects with severe cardiovascular disease;

   1. New York Heart Association (NYHA) Stage III or IV congestive heart failure;
   2. episode of myocardial infarction or coronary artery bypass grafting (CABG) ≤ 6 months prior to enrollment;
   3. clinically significant ventricular arrhythmia, or history of unexplained syncope, non-vasovagal or not due to dehydration;
   4. history of severe non-ischemic cardiomyopathy;
   5. reduced left ventricular ejection fraction (LVEF <55%), abnormal septal thickness and atrial size associated with myocardial amyloidosis, as assessed by echocardiography or multigated circuit exploration (MUGA) scan;
5. Organ function is in the following abnormalities:

   1. serum aspartate aminotransferase or alanine aminotransferase > 2.5*ULN; CK > *ULN; CK-MB > *ULN; TnT > 1.5*ULN;
   2. Total bilirubin > 1.5*ULN;
   3. partial thromboplastin time or activated partial thromboplastin time or international normalized ratio > 1.5*ULN in the absence of anticoagulant therapy;
6. Patients who have planned or may plan to undergo extracorporeal radiation therapy or surgery for prostate cancer during the study period;
7. Prior anti-IGF-1R monotherapy and any immune checkpoint inhibitor therapy;
8. Intolerance to anti-IGF-1R monotherapy drugs and immune checkpoint inhibitors;
9. uncontrolled major active infectious disease, cardiovascular disease, pulmonary disease, hematologic disease, or psychiatric disease;
10. In the opinion of the investigator, not suitable for participation in this clinical study;

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse event incidence rate | Through primary completion of study which may take up to 6 months.
  Incidence rate of adverse events graded according to the National Cancer Institute Common Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
3-month PSA progression-free survival (PSA-PFS) | 3 months after first infusion
  Time from enrollment to PSA progression as defined by PCWG3 or patient death.
6-month imaging progression-free survival (rPFS): | 6 months after first infusion
  Time from enrollment to imaging progression or death from any cause, to be evaluated in conjunction with the RECIST 1.1 criteria and the PCWG3 criteria.
6-month PSA progression-free survival (PSA-PFS) | 6 months after first infusion
  Time from enrollment to PSA progression as defined by PCWG3 or patient death.
PSA Response Rate | Through primary completion of study which may take up to 6 months.
  Percentage of PSA decline from baseline according to PCWG3 criteria
Disease Control Rate | Through primary completion of study which may take up to 6 months.
  Defined as the proportion of patients whose tumors shrunk or remained stable for a certain period of time after treatment, judged according to RECIST 1.1 and PCWG3 to include the proportion of patients with complete remission (CR), partial remission (PR), and stable disease (SD).
Objective Response Rate | Through primary completion of study which may take up to 6 months.
  Define the proportion of patients with disease CR or PR as determined by RECIST 1.1 and PCWG3 , after treatment;
Overall Survival | Through primary completion of study which may take up to 6 months.
  Defined as the time from randomization grouping to the last available assessment or death;
Incidence of bone metastasis-related events (SREs) | Through primary completion of study which may take up to 6 months.
  Incidence of bone radiotherapy (including radioisotopes), pathologic fractures (excluding trauma), spinal cord compression, and bone surgery.
Quality of life (QoL) | Through primary completion of study which may take up to 6 months.
  QoL was monitored using the validated and self-rated EORTCQLQ-C30
Quality of life (QoL) FACT-P questionnaire | Through primary completion of study which may take up to 6 months.
  QoL was monitored using the validated and self-rated questionnaire
Time to pain progression | Through primary completion of study which may take up to 6 months.
  Time from the date of randomization to the date on which the pain severity score (using the BPI-SF) increased by 30% or more from baseline. Or the time from the date of randomization to the date of observation of a 2-point increase from baseline in the BPI-SF worst pain intensity (point 3 on the scale) on 2 consecutive assessments ≥4 weeks apart or initiation of chronic opioid use, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Shancheng Ren, MD,PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the consent and approval of principal investigator, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 1 year after the publication of results
Access Criteria: Information regarding submitting proposals and accessing data maybe requested from the principal investigator by e-mail.